CLINICAL TRIAL: NCT06588634
Title: The PERSEVERE Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inari Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-002
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Pulmonary Embolism; Pulmonary Thromboembolism
Keywords: PE; Pulmonary Embolism; FlowTriever; CDT; Catheter Directed Thrombolysis; Anticoagulation
MeSH Terms: conditions — Pulmonary Embolism | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- FlowTriever (Active Comparator)
  Interventions: Device: FlowTriever System
- Standard of Care (Active Comparator)
  Interventions: Procedure: Standard of Care

INTERVENTIONS:
Device: FlowTriever System — Mechanical thrombectomy for pulmonary embolism
  Arms: FlowTriever
Procedure: Standard of Care — Standard of care treatment for pulmonary embolism
  Arms: Standard of Care

SUMMARY:
Randomized Controlled Trial of High-Risk Pulmonary Embolism Comparing FlowTriever System vs. Standard of Care

ELIGIBILITY:
Inclusion Criteria:

1. Age at enrollment ≥18 years
2. Objective evidence of a proximal filling defect in at least one main or lobar pulmonary artery
3. High-risk class of acute PE
4. RV dysfunction, as defined RV/LV ratio ≥1.0
5. Willing and able to provide informed consent, or if unable, through a Legal Authorized Representative, with permitting research without prior consent as a third option (for Europe and UK sites only), provided compliance with IRB/EC approvals and adherence to regulatory, ethical and national standards

Exclusion Criteria:

1. Prolonged cardiac arrest with loss of consciousness associated with neurological deficit.
2. Imaging evidence or other evidence that suggests, in the opinion of the Investigator, the patient is not appropriate for catheter-based intervention
3. Known pre-existing CTEPH, or CT signs of chronic PE that may point to pre-existing CTEPH
4. Recent stroke (<14 days)
5. Recent cranial or spinal surgery (<14 days)
6. Life-threatening active bleeding or hemorrhage into a critical area
7. Known intracranial tumor
8. End-stage medical condition with life expectancy <3 months (irrespective of the severity of acute PE), as determined by the Investigator
9. Known sensitivity to radiographic contrast agents that, in the Investigator's opinion, cannot be adequately pre-treated
10. Inability to anticoagulate the patient, or known to have heparin-induced thrombocytopenia (HIT)
11. Current participation in another drug or device study that may interfere with the conduct of this trial
12. Ventricular arrhythmias refractory to treatment at the time of enrollment
13. Subject has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the subject (e.g., compromise the well-being or that could prevent, limit, or confound the protocol-specified assessments), including a contraindication to use of FlowTriever System per local approved labeling
14. Subject is part of a vulnerable population (e.g., currently pregnant, breastfeeding or incarcerated) per local definitions
15. Subject was previously enrolled in this study
16. Subject has received prior thrombolytic (systemic or catheter-directed) therapy for any reason or thrombectomy (surgical or catheter-based) therapy for index PE, within 30 days prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Composite clinical endpoint of the following adjudicated events: | The earlier of initial hospital discharge or 7 days after randomization
  1. All-cause mortality
  2. Cardiac arrest
  3. Bailout to an alternative therapeutic strategy
  4. Major bleeding
  5. ECMO life support

SECONDARY OUTCOMES:
All-cause mortality | At the earlier of initial hospital discharge or 7 days post randomization and at 3-month visit
Cardiac arrest | At the earlier of initial hospital discharge or 7 days post randomization
Bailout to an alternative therapeutic strategy | At the earlier of initial hospital discharge or 7 days post randomization
Major bleeding | At the earlier of initial hospital discharge or 7 days post randomization and at 3-month visit
ECMO life support | 7 days post-randomization
PE-related mortality | 3 months
All-cause and PE-related readmissions | 30 days and 90 days
Days alive outside hospital | 90 days
PE-related quality of life, by PEmb-QoL | 3 months
General health-related quality of life, by EQ-5D-5L | 3 months
Post-PE Impairment diagnosis | 3 months
Change in the RV/LV diastolic diameter ratio (RV/LV) as measured by echocardiography from baseline | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Meneveau, MD PhD, Principal Investigator — Centre Hospitalier Universitaire Hôpital Jean Minjoz, Besançon, France; Stavros Konstantinides, MD PhD, Principal Investigator — Center for Thrombosis and Hemostasis, University Medical Center of the Johannes Gutenberg-University Mainz, Germany; John M Moriarty, MD, Principal Investigator — Westwood Imaging Center & Interventional Radiology Clinic - UCLA, CA, USA; Jay Giri, MD, MPH, Principal Investigator — Penn Medicine, Philadelphia, PA, USA
Locations (25):
- United States (12):
  - Yale University, New Haven, Connecticut
  - Orlando Health Regional Medical Center, Orlando, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Emory University, Atlanta, Georgia
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Northwell Health, Bay Shore, New York
  - SUNY, The University at Buffalo, Buffalo, New York
  - UPHS Penn Health System, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - HCA Tristar/Centennial, Nashville, Tennessee
  - HCA Medical City Heart & Spine, Dallas, Texas
  - HCA Methodist Health San Antonio, San Antonio, Texas
- France (4):
  - Besançon University Hospital, Besançon
  - Hopital Arnaud de Villeneuve, Montpellier, Montpellier
  - CHU Nîmes Caremeau, Nîmes
  - Hôpital Européen Georges-Pompidou, Paris, Paris
- Germany (5):
  - Klinikum Chemnitz, Chemnitz
  - Universitätsklinikum Carl Gustav Carus an der TU Dresden, Dresden
  - Universitätsmedizin Mainz, Mainz
  - Munich LMU, München
  - Universitätsklinik Regensburg, Regensburg
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona
  - Hospital Universitario La Paz Madrid, Madrid
- University Hospital Basel, Basel, Switzerland
- Royal Free Hospital London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chopard R, Hobohm L, Barco S, Bangalore S, Giri J, Mahfoud F, Moriarty J, Rosenkranz S, Sharp A, Thiele H, Toma C, Tapson VF, Markovitz CD, Rosenberg SP, Konstantinides S, Meneveau N. Large-bore mechanical thrombectomy vs standard of care for acute high-risk pulmonary embolism: Rationale and design of the PERSEVERE randomized controlled trial. Am Heart J. 2025 Dec 24;294:107331. doi: 10.1016/j.ahj.2025.107331. Online ahead of print. PMID 41453591